CLINICAL TRIAL: NCT05406882
Title: The Effects of Bifidobacterium and Lactobacillus Tablets Combined With Compound Glutamine in the Prevention and Treatment of Radiation Proctitis.
Brief Title: The Effects of Probiotics Combined With Glutamine in the Prevention and Treatment of Radiation Proctitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wang Xin, Professor, West China Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HX-H2112345
Record Dates: First submitted 2022-05-06; First posted 2022-06-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Radiation Proctitis; Probiotics; Glutamine; Gut Microbiota; Bifidobacterium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination therapy group (Experimental): From the first day of chemoradiotherapy, live combined Bifidobacterium and Lactobacillus tablets(2000mg each time, 3 times/day) combined with compound glutamine enteric-coated capsules (3 capsules each time, 3 times/day) until 1 month after the end of chemoradiotherapy.
  Interventions: Drug: Live Combined Bifidobacterium and Lactobacillus Tablets、Compound Glutamine Entersoluble capsules
- control group (No Intervention): After the start of chemoradiotherapy, the control group don't take the experimental drug orally . When patients have radiation proctitis of grade ≥2, they would be crossed over to the combined treatment group：live combined Bifidobacterium and Lactobacillus tablets(2000mg each time, 3 times/day) combined with compound glutamine enteric-coated capsules (3 capsules each time, 3 times/day) until 1 month after the end of chemoradiotherapy.

INTERVENTIONS:
Drug: Live Combined Bifidobacterium and Lactobacillus Tablets、Compound Glutamine Entersoluble capsules — Live Combined Bifidobacterium and Lactobacillus Tablets：probiotics. Compound Glutamine Entersoluble capsules：combined traditional Chinese medicine and glutamine
  Other Names: Probiotics、Glutamine
  Arms: combination therapy group

SUMMARY:
Radiation proctitis is a common complication after radiation therapy for pelvic tumors. The investigators found that live bifidobacterium and lactobacillus tablets combined with compound glutamine enteric-coated capsules can significantly relieve the symptoms of radiation proctitis through preliminary clinical practice, but the mechanism is unknown. Through a prospective randomized controlled study, this study intends to investigate the incidence of grade 2 or higher acute radiation proctitis in patients of locally advanced rectal cancer after radiotherapy with the combined therapy. And through various scales, next-generation sequencing methods and other methods to evaluate the clinical symptoms, colonoscopy, imaging, and changes in the species and abundance of intestinal flora before and after treatment. To further explore the related pathways and mechanisms affecting radiation proctitis.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced rectal adenocarcinoma diagnosed by histopathology; clinical stage T3/4 or N+(AJCC,8th), no metastasis; and planned to receive preoperative neoadjuvant concurrent chemoradiotherapy.
* without other malignant tumors;
* Those without serious heart, liver, kidney and other diseases;
* ECOG score: 0-1.

Exclusion Criteria:

* Complicated with ulcerative colitis or Crohn's disease;
* Complicated with severe organ insufficiency, severe diabetes, and heart disease;
* Pregnant and lactating women;
* Abnormal bowel movements with systemic and metabolic diseases;
* The patient has a history of using systemic antibiotics and intestinal active bacteria in the past 1 month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation proctitis | two months
  Incidence of grade ≥2 radiation proctitis in combination therapy group

SECONDARY OUTCOMES:
remission rate of radiation proctitis | two months
  remission rate of radiation proctitis after combined treatment in control group developed radiation proctitis of grade ≥2

OTHER OUTCOMES:
Evaluation of radiation proctitis by LENT SOMA Score | two months
  Evaluation of radiation proctitis with clinical symptoms using LENT SOMA Score.The minimum value is 0, and maximum is 4. Higher scores mean a worse outcome.
Evaluation of radiation proctitis by rectal chemoradiotherapy toxicity scale | two months
  Evaluation of radiation proctitis with clinical symptoms using rectal chemoradiotherapy toxicity scale.The minimum value is 0, and maximum is 5. Higher scores mean a worse outcome.
Evaluation of radiation proctitis by fiberoptic proctoscopy | two months
  Evaluation of radiation proctitis with fiberoptic proctoscopy using Vienna Rectoscopy Score. The minimum value is 0, and maximum is 3/4. Higher scores mean a worse outcome.
changes in gut microbiota by 16S rRNA sequencing technology | two months
  To detect changes in gut microbiota with 16S rRNA sequencing，including changes in species diversity and abundance of gut microbiota.
Changes in serum inflammatory factors | two months
  Assess changes in serum inflammatory factors , including IL-2、IL-6，CRP、TNFa, etc.
QOL C29 | two months
  Assess patients' subjective feeling of life using EORTC QOL C29.The minimum value is 1, and maximum is 4. Higher scores mean a worse outcome.
QOL C30 | two months
  Assess patients' subjective feeling of life using EORTC QOL C30.The minimum value is 1, and maximum is 4. Higher scores mean a worse outcome.
tumor imaging assessment | two months
  Evaluation of tumor changes with imaging methods，including treatment response with complete response, partial response or stable disease according to RECIST 1.1 after 1 month after concurrent chemoradiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: xin wang, Principal Investigator — China, SiChuan West China Hospital
Locations (2):
- China (2):
  - West China Hospital, Chengdu, Sichuan
  - Xin Wang, Chengdu, Sichuan